CLINICAL TRIAL: NCT07200856
Title: Impact of Nocturnal Blood Pressure Dipping on Ventricular Repolarization in Hypertensive Patients
Brief Title: Nocturnal Blood Pressure Dipping and Ventricular Repolarization in Hypertension
Acronym: NBP-DIP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Abdelwahab Hussein Ahmed, Dr, Assiut University
Other Study IDs: AUN-CARDIO-NBP-2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Blood Pressure Monitoring, Ambulatory; Circadian Rhythm; Electrocardiography; Ventricular Function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nocturnal Blood Pressure Dipping — Patients will be classified as dippers (≥10% nocturnal BP fall) or non-dippers (<10% nocturnal BP fall) based on 24-hour ambulatory blood pressure monitoring.

SUMMARY:
The primary aim is to determine whether non-dipping status is associated with adverse repolarization markers and impaired myocardial mechanics compared to dipper hypertensive patients. Secondary analyses will compare these findings among resistant vs. non-resistant and controlled vs. uncontrolled hypertensive groups. This study may provide new insights into the prognostic significance of blood pressure dipping patterns in hypertensive patients.

DETAILED DESCRIPTION:
Hypertension is a highly prevalent chronic condition and one of the leading causes of cardiovascular disease worldwide. It is associated with structural and electrical remodeling of the heart, including left ventricular hypertrophy, myocardial fibrosis, and impaired ventricular repolarization. These changes predispose patients to arrhythmias and adverse cardiovascular outcomes.

A physiological decline in blood pressure during nighttime, known as nocturnal dipping, represents a normal circadian rhythm and is considered a favorable prognostic sign. However, many hypertensive patients fail to show this nocturnal decline (non-dippers), which may indicate heightened sympathetic activity, impaired recovery during sleep, and increased cardiovascular risk. Identifying the impact of dipping status on cardiac electrical and mechanical function could therefore have important clinical value.

This study is designed as an observational prospective registry enrolling adult patients with essential hypertension. All participants will undergo 24-hour ambulatory blood pressure monitoring to determine dipping pattern, standard 12-lead electrocardiography for analysis of repolarization markers such as QTc, QT dispersion, and Tp-Te interval, and comprehensive transthoracic echocardiography including strain imaging to assess myocardial mechanics. Laboratory tests including electrolytes and renal function will also be performed to exclude confounding factors.

The primary objective is to evaluate the effect of nocturnal blood pressure dipping on ventricular repolarization parameters and echocardiographic findings in hypertensive patients. Secondary objectives include assessing differences between resistant and non-resistant hypertension as well as controlled and uncontrolled hypertension groups. The study is expected to provide novel insights into the prognostic role of dipping status and its association with electrical and functional cardiac abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Diagnosed with essential hypertension
* Completed 24-hour ambulatory blood pressure monitoring (ABPM)
* Availability of good-quality 12-lead ECG
* Availability of good-quality transthoracic echocardiography

Exclusion Criteria:

* Body mass index (BMI) > 34.9 kg/m²
* Atrial fibrillation or atrial flutter
* Use of QT-prolonging medications
* End-stage renal disease or liver failure
* Bundle branch block or presence of pacemaker
* Prior coronary revascularization (PCI or CABG)
* Significant electrolyte imbalance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with essential hypertension attending the Cardiology Department at Assiut University Heart Hospital. All participants will undergo 24-hour ambulatory blood pressure monitoring, electrocardiography, and echocardiography to classify them into dipper and non-dipper groups
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Effect of nocturnal BP dipping on ECG markers of ventricular repolarization | At enrollment
  Evaluation of QTc, QT dispersion, and Tp-Te interval in dipper vs. non-dipper hypertensive patients, correlated with echocardiographic changes

SECONDARY OUTCOMES:
Repolarization and echocardiographic changes in resistant vs. non-resistant hypertension | At enrollment
  Comparison of ECG and echocardiographic markers between resistant and non-resistant hypertensive groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Aboel-Kassem Farghal Abdelmegid, Study Chair — Cardiology Department - Assiut University; Noha Mohamed Gamal Hashem, Study Chair — Cardiology Department - Assiut University

REFERENCES:
- [Background] Demir M, Uyan U. Evaluation of Tp-e interval and Tp-e/QT ratio in patients with non-dipper hypertension. Clin Exp Hypertens. 2014;36(5):285-8. doi: 10.3109/10641963.2013.810233. Epub 2013 Jul 12. PMID 23848271
- [Background] Cuspidi C, Sala C, et al. Nocturnal blood pressure fall and left ventricular hypertrophy in untreated hypertensive patients. J Hypertens. 2013;31(6):1143-50.
- [Background] Morris DA, et al. Left atrial strain predicts diastolic dysfunction severity. J Am Soc Echocardiogr. 2015;28(5):556-64.
- [Background] Dudenbostel T, Calhoun DA. Resistant hypertension, left ventricular hypertrophy, and ECG changes. Curr Hypertens Rep. 2017;19(6):48.
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Goulart MA, Moreira DAR, Cesena FY, Souza JB, Laurinavicius AG, Consolim-Colombo FM, Sousa MG. Analysis of Ventricular Repolarization in Hypertensive Patients: Influence of Nocturnal Blood Pressure Dipping. Arq Bras Cardiol. 2025 Apr;122(4):e20240725. doi: 10.36660/abc.20240725. English, Portuguese. PMID 40396865